PRINCIPAL INVESTIGATOR: Hoyoung Maeng, M.D.

STUDY TITLE: A Pilot Study of Long-Term TARP Vaccination Using a

Multi-Epitope TARP Peptide Autologous Dendritic Cell Vaccination in Previously Vaccinated Men on NCI 09-C-

0139

STUDY SITE: NIH Clinical Center

Cohort: Affected Participant
Consent Version: 10/17/2019

#### WHO DO YOU CONTACT ABOUT THIS STUDY?

**Principal Investigator:** Hoyoung Maeng, MD

240-781-3253

hoyoung.maeng@nih.gov

This consent form describes a research study and is designed to help you decide if you would like to be a part of the research study.

You are being asked to take part in a research study at the National Institutes of Health (NIH). Members of the study team will talk with you about the information described in this document. Some people have personal, religious, or ethical beliefs that may limit the kinds of medical or research treatments they would want to receive (such as blood transfusions). Take the time needed to ask any questions and discuss this study with NIH staff, and with your family, friends, and personal health care providers. Taking part in research at the NIH is your choice.

If the individual being asked to participate in this research study is not able to give consent to be in this study, you are being asked to give permission for this person as their decision-maker. The term "you" refers to you as the decision-maker and/or the individual being asked to participate in this research, throughout the remainder of this document.

#### IT IS YOUR CHOICE TO TAKE PART IN THE STUDY

You may choose not to take part in this study for any reason. If you join this study, you may change your mind and stop participating in the study at any time and for any reason. In either case, you will not lose any benefits to which you are otherwise entitled. However, to be seen at the NIH, you must be taking part in a study or are being considered for a study. If you do choose to leave the study, please inform your study team to ensure a safe withdrawal from the research.

## WHY IS THIS STUDY BEING DONE?

There are not a lot of studies or literature available regarding the long-term safety of repeated peptide vaccinations in patients over a period of time. Long term vaccination may be necessary to maintain anti-tumor activity and control.

#### PATIENT IDENTIFICATION

**Consent to Participate in a Clinical Research Study** 

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)

Version Date: 10/17/2019


You were enrolled on the first-generation TARP Peptide Vaccine Study 09-C-0139 and received at least five TARP peptide Vaccine injections. You are being invited to participate in a second-generation TARP peptide vaccine study so that we can further assess the long term safety of repeated peptide vaccines and determine if the second generation ME TARP vaccine results in a greater variety and different types of immune responses.

The second-generation TARP peptide vaccine is a Multi-Epitope (ME) TARP vaccine. It is different than the first-generation TARP vaccine which was manufactured using only two peptides. The ME-Epitope TARP vaccine has the original the two peptides but also includes five new peptides for a total of seven peptides that cover the entire TARP protein. As a participant in the first-generation TARP study you will provide a unique opportunity for us to assess the impact of re-vaccination on boosting and sustaining immune responses to TARP.

Your participation in this second-generation TARP peptide vaccine study will allow us to:

- 1. Assess the long-term safety of repeated TARP peptide vaccinations. Since you have already received two years of TARP peptide immunizations, we already have two years of data already collected.
- 2. Study your immune responses to the second generation ME TARP vaccine and compare them your immune responses to the first-generation TARP vaccine on protocol 09-C-0139.

#### HOW MANY PEOPLE WILL TAKE PART IN THIS STUDY?

We would like to enroll as many of the same 40 participants that were enrolled on the first-generation TARP vaccine study.

#### DESCRIPTION OF RESEARCH STUDY

**Study Design**: This is an open label (open-label means that both you and your study doctor know what investigational vaccine you are receiving), non-randomized, long term pilot study of 96 weeks to assess the long-term safety of repeated TARP vaccination in patients that have already received the first-generation TARP vaccination

#### What will happen if you take part in this research study?

Before you begin the study, you will need to have the **screening examinations**, tests and diagnostic procedures to find out if you can be in the study. Some of these examinations, test or procedures may be repeated during the study to assure your safety and to assess your responses to the vaccines. Some of these screening tests may also be performed at your home institutions and forwarded to us. The examinations, tests, and procedures that are a part of the screening process include:

- Routine laboratory blood tests that examine your blood counts, urine and PSA as well as your kidney, liver and thyroid function.
- As part of this study, we will test you for infection with the human immunodeficiency virus (HIV), the virus that causes AIDS. If you are infected with HIV you will not be able to participate in this study. We will tell you what the results mean, how to find care, how to

#### PATIENT IDENTIFICATION

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)


avoid infecting others, how we report HIV infection, and the importance of informing your partners at possible risk because of your HIV infection.

- CT scan, Bone scan
- Physical exam with past medical history
- Medications you are currently taking
- Evaluation of performance status- how well you are able to do every day activities

## If you should meet all Eligibility Criteria and:

- You are not receiving and do not require active chemotherapy or radiation therapy for the treatment of your prostate cancer.
- You do not have a secondary malignancy requiring active treatment
- You do not have an active infection
- You are not on immunosuppressive therapy (such as systemic corticosteroid therapy).
- You do not have another significant or uncontrolled medical illness

## What happens next?

After you have been found eligible for the study, and all of your questions have been answered and you have signed the informed consent for this study you will be scheduled for an apheresis. Just as in the first-generation TARP, we will need to collect a large number of cells to custom make your vaccine. To ensure that we have sufficient cells these cells are collected during the apheresis procedure. A description of the apheresis procedure is below. Apheresis may be required to be repeated during study participation if not enough cells have initially been obtained.

## **Apheresis:**

The procedure for obtaining certain types of blood cells through apheresis is a very common procedure that is done routinely here in the Clinical Center with very few risks. Apheresis requires you to have a needle placed in your arm where the blood can be removed from you and circulated through a cell separator machine (a machine that divides whole blood into red cells, plasma (the serum part) and white cells (that includes lymphocytes and monocytes). The white blood cells are removed and the plasma and red cells are returned to you through another needle in your other arm. The procedure takes approximately 1 to 3 hours to complete. One of the purposes of this procedure is to allow the investigator to collect a sufficient number of immune cells to measure the immune response to the vaccine. This testing will provide no benefit to you and is part of the experimental portion of this research study. Patients do not need to be hospitalized for the procedure. The apheresis procedure will be done at the Department of Transfusion Medicine (Blood Bank) in the NIH Clinical Center and is carried out by trained nurses supervised by Blood Bank physicians.

Potential side effects associated with Apheresis: you may have some tingling in your face and lips due to the medicine used to keep your blood from clotting during the procedure. The nurses may give you calcium-containing tablets, such as TUMS; to chew that takes away this tingling. Some patients may feel faint or light-headed during or after this procedure. We ask that you make sure you have a good meal and are well hydrated prior to coming to the apheresis lab.

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)


## **During the Study**

With each clinic visit you will have a physical exam, laboratory and research blood draws. You will be asked about any side effects or illnesses you may have had between visits. You will also be asked about your medications.

We will continue to monitor your PSA and unless you are on androgen deprivation therapy, calculate your PSA doubling time (PSADT). You will continue to monitor your injection site and bring your Vaccine Report Card to your visits.

#### **Birth Control**

If you are the partner of a woman who can become pregnant, you will need to practice an effective form of birth control before starting study treatment, during study treatment and for 30 days after your last dose of vaccine. If you think your partner is pregnant, you should tell your study doctor or nurse at once.

Effective forms of birth control include:

- abstinence
- vasectomy

#### RISKS OR DISCOMFORTS OF PARTICIPATION

## What side effects or risks can I expect from being in this study?

Everyone taking part in the study will be monitored very carefully for any side effects and we will ask you to fill out a Vaccine Report Card to monitor any symptoms you may have following your vaccine injection. Since we don't know all the side effects that may be associated with these vaccines, it is very important that you report any changes that you may notice, even if your study team does not specifically ask about them.

In the first generation TARP vaccine study, the most commonly reported side effects were local injection site reactions such as pain, soreness, swelling, itching and /or redness at the site where the vaccine was given. The second generation ME TARP vaccine being investigated in this study may result in stronger or different types of immune responses that may have unexpected and unknown side effects such as:

- Fever
- Chills
- Rash
- Flu-like symptoms
- Headache

It is also possible that you could develop an immune response to the ME TARP vaccine that will cause inflammation in your prostate gland or other organs such as your thyroid. However these problems were not observed with the first generation TARP vaccine and we will be monitoring you closely for them.

In general, peptide vaccines that have been given to cancer patients have been found to be safe and very well tolerated.

#### PATIENT IDENTIFICATION

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)


#### Likely

• Injection site reactions, including possible pain or soreness, swelling, itching and/or redness at the injection site.

## POTENTIAL BENEFITS OF PARTICIPATION

Taking part in this study may or may not provide a direct benefit to you. It is unknown whether vaccination with ME-TARP DCs will stimulate an immune response by your body.

If ME-TARP DC vaccination stimulates an immune response that slows how fast your PSA is rising, it may help your body to fight your prostate cancer more effectively. Since this is an experimental therapy, no benefit can be promised. However, the information we obtain from both the laboratory studies, long term safety and your response to ME TARP vaccination may also allow us to understand and better treat cancer for future patients.

#### ALTERNATIVE APPROACHES OR TREATMENTS

## What other choices do I have if I do not take part in this study?

## For Patients That Have Stage D0 Disease at the Time of Enrollment

Treatment options for patients with elevated PSA levels but no evidence of disease spread to other organs following primary treatment for their prostate cancer (Stage D0) includes watchful waiting or androgen deprivation hormone therapy. However, it is unclear for patients with this stage of disease what the best approach is. Because many patients prefer to avoid the side effects of hormonal treatment (impotence, hot flashes, loss of libido, breast tenderness, osteoporosis and bone fractures) watchful waiting is often chosen.

If you develop evidence of disease progression, involving spread of your prostate cancer to the bone, brain or other organs, alternative treatments/therapy for your cancer may include:

- ➤ Getting treatment or care for your cancer without being in a study. Some examples include: treatment with hormone therapy, radiotherapy, chemotherapy or a combination of these approaches.
- ➤ Getting comfort care, also called palliative care. This type of care helps reduce pain, tiredness, appetite problems and other problems caused by the cancer. It does not treat the cancer directly. Instead, it tries to improve how you feel. Comfort care tries to keep you as active and comfortable as possible.
- Taking part in another study. No further therapy at all

If you choose to receive hormone therapy treatment through your local doctor you will be allowed to remain on study so that we can continue to monitor you for safety and for your immune responses to the TARP vaccine. If you require active treatment with chemotherapy or radiotherapy for your prostate cancer you will be taken off the study.

# For Patients That Have Documented Locally Recurrent or Metastatic Disease at the Time of Enrollment

If you have previously documented locally recurrent or metastatic prostate cancer when you enroll in this study, you will be allowed to receive (or continue receiving) hormone therapy through your

## PATIENT IDENTIFICATION

**Consent to Participate in a Clinical Research Study** 

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)


local oncologist. However, if you have further disease progression while on this protocol that requires you to get active chemotherapy or radiation therapy for your prostate cancer, you will be taken off the study.

Each of these alternative therapies has a unique set of benefits and risks. Your physician will discuss these options with you. Furthermore, other centers are performing clinical trials with investigational agents including immune-based therapies and vaccines as well as standard chemotherapy that you may want to consider as an alternative to this proposed trial.

#### STOPPING THERAPY

Your doctor may decide to stop your therapy for the following reasons:

- if he/she has repeated problems creating a vaccine that meets NIH standards from your cells
- if your vaccine is delayed for more than 6 weeks
- if your disease spreads to other parts of your body (D0 patients only)
- if your PSADT falls below 3 months or is reduced by more than half of what it was before you began the study (D0 patients only)
- if your prostate disease worsens and you require chemotherapy or radiation
- if your treatment is delayed more than 6 weeks
- if you develop another cancer during the course of the study
- if he/she believes that it is in your best interest
- if he/she decides to end the study

You can stop taking part in the study at any time. However, if you decide to stop taking part in the study, we would like you to talk to the study doctor and your regular doctor first

If you decide at any time to withdraw your consent to participate in the trial, we will not collect any additional medical information about you. If you withdraw your consent and leave the trial, any samples of yours that have been obtained for the study and stored at the NCI can be destroyed upon request. However, any samples and data generated from the samples that have already been distributed to other researchers or placed in the research databases cannot be recalled and destroyed. Research Subject's Rights

Participation in this research study is voluntary. You will get a copy of this Informed Consent and you may withdraw your consent to participate at any time. There are no penalties for leaving the study. Patients may ask our staff to answer any and all questions and we invite you to do so.

## **CONFLICT OF INTEREST**

The National Institutes of Health (NIH) reviews NIH staff researchers at least yearly for conflicts of interest. This process is detailed in a Protocol Review Guide. You may ask your research team for a copy of the Protocol Review Guide or for more information. Members of the research team who do not work for NIH are expected to follow these guidelines but they do not need to report their personal finances to the NIH.

#### PATIENT IDENTIFICATION

**Consent to Participate in a Clinical Research Study** 

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)


Members of the research team working on this study may have up to \$15,000 of stock in the companies that make products used in this study. This is allowed under federal rules and is not a conflict of interest.

The National Institutes of Health and the research team for this study have developed a vaccine being used in this study. This means it is possible that the results of this study could lead to payments to NIH scientists and to the NIH. By law, government scientists are required to receive such payments for their inventions. You will not receive any money from the development of multi-epitope TARP peptide vaccine.

The National Institutes of Health and the research team for this study are working in collaboration with PDS Biotechnology and with RareCyte, Inc. to perform tests on your samples. The companies also provides financial support for this study.

#### USE OF SPECIMENS AND DATA FOR FUTURE RESEARCH

To advance science, it is helpful for researchers to share information they get from studying human samples. They do this by putting it into one or more scientific databases, where it is stored along with information from other studies. A researcher who wants to study the information must apply to the database and be approved. Researchers use specimens and data stored in scientific databases to advance science and learn about health and disease.

We plan to keep some of your specimens and data that we collect and use them for future research and share them with other researchers. We will not contact you to ask about each of these future uses. These specimens and data will be stripped of identifiers such as name, address or account number, so that they may be used for future research on any topic and shared broadly for research purposes. Your specimens and data will be used for research purposes only and will not benefit you. It is also possible that the stored specimens and data may never be used. Results of research done on your specimens and data will not be available to you or your doctor. It might help people who have cancer and other diseases in the future.

If you do not want your stored specimens and data used for future research, please contact us in writing and let us know that you do not want us to use your specimens and/or data. Then any specimens that have not already been used or shared will be destroyed and your data will not be used for future research. However, it may not be possible to withdraw or delete materials or data once they have been shared with other researchers.

## COMPENSATION, REIMBURSEMENT, AND PAYMENT

## Will you receive compensation for participation in the study?

Some NIH Clinical Center studies offer compensation for participation in research. The amount of compensation, if any, is guided by NIH policies and guidelines.

You will not receive compensation for participation in this study.

## Will you receive reimbursement or direct payment by NIH as part of your participation?

Some NIH Clinical Center studies offer reimbursement or payment for travel, lodging or meals while participating in the research. The amount, if any, is guided by NIH policies and guidelines.

On this study, the NCI will cover the cost for some of your expenses. Some of these costs may be paid directly by the NIH and some may be reimbursed after you have paid. Someone will work with you to provide more information.

## Will taking part in this research study cost you anything?

NIH does not bill health insurance companies or participants for any research or related clinical care that you receive at the NIH Clinical Center.

- If some tests and procedures performed outside the NIH Clinical Center, you
  may have to pay for these costs if they are not covered by your insurance
  company.
- Medicines that are not part of the study treatment will not be provided or paid for by the NIH Clinical Center.
- Once you have completed taking part in the study, medical care will no longer be provided by the NIH Clinical Center.

#### CLINICAL TRIAL REGISTRATION AND RESULTS REPORTING

A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

## CONFIDENTIALITY PROTECTIONS PROVIDED IN THIS STUDY

## Will your medical information be kept private?

We will do our best to make sure that the personal information in your medical record will be kept private. However, we cannot guarantee total privacy. Organizations that may look at and/or copy your medical records for research, quality assurance, and data analysis include:

- The NIH and other government agencies, like the Food and Drug Administration (FDA), which are involved in keeping research safe for people.
- National Institutes of Health Intramural Institutional Review Board
- The study Sponsor Center for Cancer Research or their agents.
- Qualified representatives from RareCyte, Inc., companies that will supply agents used to perform studies on your cells.

When results of an NIH research study are reported in medical journals or at scientific meetings, the people who take part are not named and identified. In most cases, the NIH will not release any information about your research involvement without your written permission. However, if you sign a release of information form, for example, for an insurance company, the NIH will give the

#### PATIENT IDENTIFICATION

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)


insurance company information from your medical record. This information might affect (either favorably or unfavorably) the willingness of the insurance company to sell you insurance.

If we share your specimens or data with other researchers, in most circumstances we will remove your identifiers before sharing your specimens or data. You should be aware that there is a slight possibility that someone could figure out the information is about you.

Further, the information collected for this study is protected by NIH under a Certificate of Confidentiality and the Privacy Act.

## **Certificate of Confidentiality**

To help us protect your privacy, the NIH Intramural Program has received a Certificate of Confidentiality (Certificate). With this certificate, researchers may not release or use data or information about you except in certain circumstances.

NIH researchers must not share information that may identify you in any federal, state, or local civil, criminal, administrative, legislative, or other proceedings, for example, if requested by a court.

The Certificate does not protect your information when it:

- 1. is disclosed to people connected with the research, for example, information may be used for auditing or program evaluation internally by the NIH; or
- 2. is required to be disclosed by Federal, State, or local laws, for example, when information must be disclosed to meet the legal requirements of the federal Food and Drug Administration (FDA);
- 3. is for other research;
- 4. is disclosed with your consent.

The Certificate does not prevent you from voluntarily releasing information about yourself or your involvement in this research.

The Certificate will not be used to prevent disclosure to state or local authorities of harm to self or others including, for example, child abuse and neglect, and by signing below you consent to those disclosures. Other permissions for release may be made by signing NIH forms, such as the Notice and Acknowledgement of Information Practices consent.

## **Privacy Act**

The Federal Privacy Act generally protects the confidentiality of your NIH medical records we collect under the authority of the Public Health Service Act. In some cases, the Privacy Act protections differ from the Certificate of Confidentiality. For example, sometimes the Privacy Act allows release of information from your medical record without your permission, for example, if it is requested by Congress. Information may also be released for certain research purposes with due consideration and protection, to those engaged by the agency for research purposes, to certain federal and state agencies, for HIV partner notification, for infectious disease or abuse or neglect reporting, to tumor registries, for quality assessment and medical audits, or when the NIH is involved in a lawsuit. However, NIH will only release information from your medical record if it is permitted by both the Certificate of Confidentiality and the Privacy Act.

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)


#### POLICY REGARDING RESEARCH-RELATED INJURIES

The NIH Clinical Center will provide short-term medical care for any injury resulting from your participation in research here. In general, no long-term medical care or financial compensation for research-related injuries will be provided by the NIH, the NIH Clinical Center, or the Federal Government. However, you have the right to pursue legal remedy if you believe that your injury justifies such action.

## PROBLEMS OR QUESTIONS

If you have any problems or questions about this study, or about your rights as a research participant, or about any research-related injury, contact the Principal Investigator, Hoyoung Maeng, MD (240-781-3253 or <a href="hoyoung.maeng@nih.gov">hoyoung.maeng@nih.gov</a>). You may also call the NIH Clinical Center Patient Representative at 301-496-2626, or the NIH Office of IRB Operations at 301-402-3713, if you have a research-related complaint or concern.

#### CONSENT DOCUMENT

Please keep a copy of this document in case you want to read it again.


# MEDICAL RECORD

## CONSENT TO PARTICIPATE IN AN NIH CLINICAL RESEARCH STUDY

| Signature of Research Participant | Print Name of Research Participa | ant Date |
|---|---|---|
| about this study and have been given the to make research decisions on behalf of the | AR) for an Adult Unable to Consent: opportunity to discuss it and to ask questine adult participant unable to consent and information in the above consent was described in the study. | ions. I am legally authorize have the authority to provid |
| Signature of LAR | Print Name of LAR | Date |
| Investigator: | | |
| Signature of Investigator | Print Name of Investigator | Date |
| Witness to the oral short-form consent short-consent process and this English cotranslation. | Print Name of Investigator process only: This section is only required by the IRE | red if you are doing the ora |
| | process only: This section is only requir | red if you are doing the ora |
| Witness to the oral short-form consent short-consent process and this English cotranslation. Witness: Signature of Witness* | process only: This section is only requirement form has been approved by the IRE | red if you are doing the ora B for use as the basis of Date |
| Witness to the oral short-form consent short-consent process and this English contranslation. Witness: Signature of Witness* *NIH ADMINISTRATIVE SECTIO INTERPRETER: An interpreter, or other individual, we should not be a short-form consent short-form | Print Name of Witness | Date The USE OF A referred language facilitate |

NIH-2977 (4-17)


File in Section 4: Protocol Consent (1)